CLINICAL TRIAL: NCT07006584
Title: Impact of a Functional Gait Training Program as a Complementary Strategy to Improve Physical Function in Older Adults
Brief Title: Gait Reeducation Program in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Alberto Bermejo Franco, Principal Investigator, Clinical Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 182-2023-CIEI-FMH-USMP
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Older Adults (65 Years and Older); Balance; Gait Disorders; Physical Performance; Calf Muscle Weakness; Abdominal; Sarcopenia; Handgrip Strength; Functional Capacity
Keywords: Frailty; Aged; Mobility; Physical Performance; Healthy Aging; Physical Therapy
MeSH Terms: conditions — Mobility Limitation; Sarcopenia; Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Physical activity workshops) (Active Comparator): Group A attended only the physical activity workshops offered by Centro Integral del Adulto Mayor (CIAM), consisting of one weekly class each of gymnastics, dance, swimming, and Tai Chi, held on different days of the week.
  Interventions: Other: Active Comparator #1
- Group B (Physical activity workshops+functional gait training with SSM Fisior® program) (Experimental): Group B participated in the same workshops and additionally completed functional gait training using the SSM Fisior® program. The intervention period lasted 12 weeks for both groups, with 2 additional weeks allocated for baseline and post-intervention assessments (T1 and T2).
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — Group B participated in the same workshops and additionally completed functional gait training using the SSM Fisior® program. The intervention period lasted 12 weeks for both groups, with 2 additional weeks allocated for baseline and post-intervention assessments (T1 and T2).
  Arms: Group B (Physical activity workshops+functional gait training with SSM Fisior® program)
Other: Active Comparator #1 — Group A attended only the physical activity workshops offered by Centro Integral del Adulto Mayor (CIAM), consisting of one weekly class each of gymnastics, dance, swimming, and Tai Chi, held on different days of the week.
  Arms: Group A (Physical activity workshops)

SUMMARY:
The sequential square mat (SSM) Fisior® program is a novel functional gait training tool designed to enhance motor control, coordination, and strength through guided step sequences on a visual-tactile platform. The objective of the present study is to evaluate the effects of incorporating the SSM Fisior® gait training program into routine physical activity workshops for older adults. Specifically, the study aims to assess its impact on skeletal muscle quantity, strength, and performance, as well as overall functional capacity, in a population of older adults attending a municipal community center (Centro Integral del Adulto Mayor, CIAM) in Lima, Peru.

DETAILED DESCRIPTION:
The present study is a randomized was carried out with adults aged 60 years and older recruited from the Comprehensive Center for Older Adults (CIAM) in the Lince district of Lima, Peru. The study adhered to the ethical principles outlined in the Declaration of Helsinki, and its protocol (182-2023-CIEI-FMH-USMP) received approval from the Institutional Ethics Committee of the Faculty of Human Medicine at the University of San Martín de Porres (USMP), Lima, Peru.

Participants were eligible if they were 60 years or older, were not institutionalized, scored 24 or higher on the Mini-Mental State Examination (MMSE), indicating no cognitive impairment, could communicate effectively, were able to stand up and walk at least 10 meters unassisted, scored 60 or higher on the Barthel Index (indicating sufficient functional independence). Furthermore, participants were excluded if they had a medical condition that contraindicated gait training and exhibited severe cognitive or behavioral impairments that would prevent them from completing the training program.

A simple randomization process was used to assign participants to two groups: Group A and Group B. The randomization was performed using a computer-generated random number sequence with Microsoft Excel, and it was conducted after participant enrollment to ensure allocation concealment. Group A attended only the physical activity workshops offered by Centro Integral del Adulto Mayor (CIAM), consisting of one weekly class each of gymnastics, dance, swimming, and Tai Chi, held on different days of the week. Group B participated in the same workshops and additionally completed functional gait training using the SSM Fisior® program. The intervention period lasted 12 weeks for both groups, with 2 additional weeks allocated for baseline and post-intervention assessments (T1 and T2). All assessments and activities were carried out at the CIAM center in Lince (Lima, Peru), between October and December 2023.

ELIGIBILITY:
Inclusion Criteria:

They where elegible if they were:

* 60 years or older.
* Not institutionalized.
* Scored 24 or higher on the Mini-Mental State Examination (MMSE), indicating no cognitive impairment.
* Could communicate effectively.
* Able to stand up and walk at least 10 meters unassisted
* Scored 60 or higher on the Barthel Index (indicating sufficient functional independence).

Exclusion Criteria:

Furthermore, participants were excluded if they:

* Had a medical condition that contraindicated gait training and exhibited severe cognitive or behavioral impairments that would prevent them from completing the training program.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Physical Performance | Baseline and Week 12
  Several tools have been proposed to evaluate mobility and to assess it. In this study, physical performance was measured using the Short Physical Performance Battery (SPPB), which has been validated for use in older populations. This test includes three components: balance (foot together, semi-tandem, tandem), 4-meter gait speed, and chair stand test (standing and sitting five times). The SPPB scores each timed task based on predefined thresholds, resulting in a total score ranging from 0 (worst performance) to 12 (best performance).
  The SPPB was designed to quickly identify the physical status of older adults by assessing lower limb functionality. Performance in these tests is strongly associated with mobility-related disability and serves as an independent predictor of short-term mortality and institutionalization. The medical community uses SPPB, among other tools, as a primary approach to detect and identifying frailty.

SECONDARY OUTCOMES:
Gait Speed | Baseline and Week 12
  Gait speed was assessed using the Timed Up and Go Test (Up&Go), a fundamental mobility indicator. This test measures the time taken for a person to rise from a chair with armrests, walk 3 meters, return, and sit back down.
Calf Circumference | Baseline and Week 12
  This standardized approach ensured reliability and accuracy in the calf circumference data, strengthening its role as a valid anthropometric marker for evaluating nutritional and functional health status in older adults.
Abdominal Circumference | Baseline and Week 12
  Abdominal circumference (AC), also referred to as waist circumference, is an important anthropometric parameter commonly used to assess nutritional status and central adiposity. It is a well-established indicator of cardiometabolic risk, strongly associated with conditions such as cardiovascular and cerebrovascular disease.
  In this study, AC was measured following standard anthropometric procedures, specifically 2.5 cm above the navel, using a non-elastic, flexible measuring tape. Participants were instructed to stand upright with feet shoulder-width apart, arms relaxed at their sides, and abdomen relaxed but not contracted. The measurement was taken at the end of a normal expiration to avoid variability caused by breathing.
  All measurements were conducted by trained health professionals experienced in anthropometric assessment. Each measurement was taken twice; if the two values differed by more than 1.0 cm, a third measurement was performed.
SARC-F (Strength, Ambulation, Rising from a chair, Stair climbing and history of Falling) | Baseline and Week 12
  SARC-F (Strength, Ambulation, Rising from a chair, Stair climbing and history of Falling) is a self-reported screening tool used in the sarcopenia diagnosis process that has been proposed and validated for various English-speaking and Latin populations. The test is based on the following questions: Ability to carry 4.5 kg; Need for assistance to cross a room; Ability to stand up from a chair; Ability to climb 10 steps; Number of falls in the past year. For the first four questions, the responses are scored as follows: None = 0, Some = 1, Much or Cannot = 2. For the fifth question, responses are scored as follows: None = 0, 1-3 falls = 1, 4 or more falls = 2. A SARC-F (Strength, Ambulation, Rising from a chair, Stair climbing and history of Falling) score > 4 indicates a positive risk for diagnosing sarcopenia.
Handgrip Strength | Baseline and Week 12
  Dynamometry, or handgrip strength measurement, is used to assess the function and strength of the upper extremities. Handgrip strength was assessed using a Jamar hydraulic handheld dynamometer (Jamar, Sammons Preston, Bolingbrook, IL), a standard and validated tool for measuring isometric grip force. Each participant performed three trials with their dominant hand, with a 60-second rest between trials to prevent fatigue. Verbal encouragement was provided during each trial to ensure maximal effort. The highest value obtained from the three attempts was used for analysis. This method is widely recommended for evaluating overall muscle strength and functional capacity in older adults.
Functional Capacity: Barthel Index | Baseline and Week 12
  The Barthel Index (BI) is considered one of the most suitable tools for identifying functional limitations that impact older adults' quality of life in home and community settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Center for Older Adults (CIAM)., Lince, Lima region, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alegre-Tamariz J, Sanchez-Medina J, Runzer-Colmenares FM, Avila-Rodriguez C, Bermejo-Franco A, Parodi JF. Impact of a functional gait training program as a complementary strategy to improve physical function in older adults: a randomized clinical trial. BMC Geriatr. 2025 Oct 21;25(1):789. doi: 10.1186/s12877-025-06471-x. PMID 41120990